CLINICAL TRIAL: NCT03456570
Title: The Efficacy of Progestins in Treatment of Functional Ovarian Cyst
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, amgad magdy saber, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Progestins and ovarian cyst
Record Dates: First submitted 2018-02-16; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Functional Ovarian Cyst; Progesterone
MeSH Terms: interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- progesterone (Active Comparator): these patients will be offered Dydrogesterone 10 mg twice daily will be offered for 10 days , then they will be seen Post-menstrual or delayed menses for 1 week after treatment
  Interventions: Drug: Dydrogesterone 10 mg
- placebo (Placebo Comparator): those patients will be offered placebo tablets twice daily will be offered for 10 days , then they will be seen Post-menstrual or delayed menses for 1 week after treatment
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dydrogesterone 10 mg — Dydrogesterone 10 mg twice daily
  Other Names: duphaston 10 mg
  Arms: progesterone
Drug: Placebo Oral Tablet — oral tablets twice daily
  Arms: placebo

SUMMARY:
The aim of this study is to determine whether the use of progesterone only pills has a beneficial effect over the expectant management of functional ovarian cyst or not , through a sample of female patients within the reproductive years

DETAILED DESCRIPTION:
An ovarian cyst is a common gynecological problem and is divided into 2 main categories; physiological and pathological In relative frequency, functional cysts account for about 24% of all ovarian cysts, benign cysts 70% and malignant 6% Functional cysts are the most common masses seen in the premenopausal ovary and are estimated to affect 8%-20% of reproductive-aged women

Pain or discomfort in the lower abdomen Severe pain from torsion (twisting) or rupture - Cyst rupture is characterized by sudden, sharp, unilateral pelvic pain; this can be associated with trauma, exercise, or coitus. Cyst rupture can lead to peritoneal signs, abdominal distention, and bleeding (which is usually self-limited) Discomfort with intercourse, particularly deep penetration Changes in bowel movements such as constipation Pelvic pressure causing tenesmus or urinary frequency Menstrual irregularities Precocious puberty and early menarche in young children Abdominal fullness and bloating Indigestion, heartburn, or early satiety Hyperpyrexia - This may result from some complications of ovarian cysts, such as ovarian torsion Adnexal or cervical motion tenderness In current clinical practice , gynecologists treat functional ovarian cysts with either oral Contraceptive pills or expectant management alone. we presume using progesterone only pills for treatment of functional ovarian cyst

ELIGIBILITY:
Inclusion Criteria:

* Female patients at reproductive age (18-44) Menstruating ovarian cyst (a cyst 3-10 cm in diameter, unilateral , unilocular ,clear content) BMI : patients with normal BMI (18.5-24.9) and overweight (25-29.9) included

Exclusion Criteria:

* Exclusion criteria are ovarian payhology (dermoid, endometriosis or malignancies)

Complicated cyst (rupture, torsion) Patients receiving hormonal treatment for the previous 3 cycles History of surgical removal of ovarian cyst Comorbidities like uncontrolled DM ,hypertension and tuberculosis

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
disappearance of cyst | 2 months
  ultrasound evaluation
  Post-menstrual or delayed menses for 1 week after treatment Patients will be asked about residual symptoms Then TVUS if
  1. resolved , another examination will be scheduled after 1 month post-menstrual
  2. decreasing in size , another course of treatment will be offered
  3. stationary or increasing ,patient will be offered COCs (0.15 mg levonorgestrel and 0.03 mg ethinyl estradiol)
  4. complicated ( torsion or rupture ) , patient will be subjected to surgery

CONTACTS AND LOCATIONS:
Overall Officials: amgad saber, bachelor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Grimes DA, Jones LB, Lopez LM, Schulz KF. Oral contraceptives for functional ovarian cysts. Cochrane Database Syst Rev. 2014 Apr 29;2014(4):CD006134. doi: 10.1002/14651858.CD006134.pub5. PMID 24782304
- [Background] Goh W, Bohrer J, Zalud I. Management of the adnexal mass in pregnancy. Curr Opin Obstet Gynecol. 2014 Apr;26(2):49-53. doi: 10.1097/GCO.0000000000000048. PMID 24614018